CLINICAL TRIAL: NCT03666364
Title: Magnetic Nanoparticle Sperm Separation for ICSI Cycles With Teratozoospermia and Over 35 Years Old Women Age
Brief Title: Magnetic Nanoparticle Sperm Separation for Teratozoospermia Male and Women Older Than 35 Years
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ibn Sina Hospital (Other Government)
Collaborators: Banon IVF Center Assiut, Egypt (Other)
Responsible Party: Principal Investigator, Muhammad Fawzy, IVF Lab Director, Ibn Sina Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: IbnSina-MNP
Record Dates: First submitted 2018-09-09; First posted 2018-09-11 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Sperm Injections, Intracytoplasmic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnetic nanoparticle selection for teratozoospermia (Experimental)
  Interventions: Other: Sperm preparation for ICSI
- Density gradient centrifugation for teratozoospermia (No Intervention)

INTERVENTIONS:
Other: Sperm preparation for ICSI — A new protocol for sperm preparation for ICSI cycles with teratozoospermia in over 35 years old women
  Arms: Magnetic nanoparticle selection for teratozoospermia

SUMMARY:
Women over 35 years old are likely to suffer from impaired oocyte repair capacity. Teratozoospermia is a condition reflects morphological affection of sperm. These spermatozoa would add an extra burden on the oocyte after ICSI. Whether selecting mature sperm by magnetic nanoparticle protocol would provide a more competent sperm to a likely affected oocyte would improve ICSI outcomes is the question of this research.

ELIGIBILITY:
Inclusion Criteria:

* women indicated for ICSI but with teratozoospermia

Exclusion Criteria:

* Women not failing in this group

Ages: 35 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1400 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | Twelve weeks of gestation

SECONDARY OUTCOMES:
Embryo development after ICSI | Six days of culture

CONTACTS AND LOCATIONS:
Locations (3):
- Egypt (3):
  - Qena Fertility Center, Qina, Qena Governorate
  - Banon Assiut, Asyut
  - IbnSina IVF Center, Sohag

IPD SHARING:
Plan to Share IPD: No